CLINICAL TRIAL: NCT04138459
Title: Development of Recovery Oriented Practices, Knowledge and Collaboration in a Norwegian Municipality. An Explorative Study
Brief Title: Recovery - a Collaborative Project
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College of Southeast Norway (Other)
Collaborators: Extrastiftelsen (Other)
Responsible Party: Sponsor
Other Study IDs: UCSNorway
Record Dates: First submitted 2019-02-26; First posted 2019-10-24 (Actual); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Mental Health Impairment; Substance Abuse
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Qualitative exploration: Ten community mental health service users will be interviewed with their most important mental health worker to explore how recovery orientation of services affects roles and collaboration.
  Interventions: Other: Not an interventional study. This is a qualitative, explorative study of recovery orientation of community mental health services

INTERVENTIONS:
Other: Not an interventional study. This is a qualitative, explorative study of recovery orientation of community mental health services — Explore recovery orientation of mental health services in a municipality through:
  1. Qualitative, in-depth interviews with service users and mental health professionals and
  2. Observational fieldwork

SUMMARY:
In Norway, official guidelines and policies state that recovery oriented services in the field of mental health and substance abuse services is a desirable goal.

This collaborative research project aims to provide in-depth knowledge of how recovery oriented practices and collaboration in the mental health and substance abuse services in the municipality of New Drammen develop over a three-year period.

Using qualitative methods, the main aim of the study is to explore what recovery orientation of services in mental health and substance abuse presupposes and involves related to roles, collaboration and knowledge.

To explore these issues, service users will be interviewed together with their primary mental health professional.

The study will also apply observational fieldwork in order to observe recovery oriented practices between service users and professionals and between professionals.

An advisory group consisting of people with background as service users, mental health clinicians and service leaders will contribute throughout the project.

.

ELIGIBILITY:
1. Adults who have received community mental health and / or substance abuse services for the past year or longer, due to moderate or severe mental health and / or substance abuse problems.

   Inclusion Criteria:
   * receives community mental health services due to mental health and /or substance abuse related problems
   * Above 18 years old

   Exclusion Criteria:
   * Under the age of 18
2. Mental health workers in the municipality, working in mental health and substance abuse services

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults who have received community mental health and / or substance abuse services for the past year or longer, due to moderate or severe mental health and / or substance abuse problems.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-05-30 (Actual); Primary Completion 2020-12-15 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Contribute to the knowledge base on what recovery orientation of services involves | The aims of the study will be explored through interviews and fieldwork over an anticipated period of 2 years
  The anticipated outcome is to obtain insight on how recovery orientation of mental health services affects roles, knowledge and collaboration in a Norwegian municipality.

CONTACTS AND LOCATIONS:
Overall Officials: Heidi c Kapstad, PhD, Study Chair — University of South-Eastern Norway
Locations (1):
- Trude G Klevan, Drammen, Norway

IPD SHARING:
Plan to Share IPD: No